CLINICAL TRIAL: NCT05778539
Title: Systematic Lateral Retinacular Release Does Not Reduce Post-Operative Anterior Knee Pain After Primary Total Knee Arthroplasty With Patellar Replacement
Brief Title: Lateral Retinacular Release in Total Knee Arthroplasty With Patellar Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Carlos Torrens, Clinical Professor, Hospital del Mar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/8993/I
Record Dates: First submitted 2023-02-27; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Anterior Knee Pain Syndrome
Keywords: Total knee arthroplasty; Patellar resurfacing; Lateral retinacular release; Anterior knee pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral retinacular release group (Experimental): During the implantation of a total knee arthroplasty a lateral retinacular release is performed
  Interventions: Procedure: Lateral retinacular release
- Non-release group (No Intervention): No aditional gesture in the lateral retinaculum is performed during the implantation of a total knee arthroplasty

INTERVENTIONS:
Procedure: Lateral retinacular release — During the implantation of a total knee arthroplasty a lateral retinacular release is performed in the intervention group
  Arms: Lateral retinacular release group

SUMMARY:
The aim of this study is to assess the effect of systematic lateral retinacular release on anterior knee pain, as well as its impact on the functional and radiological outcomes after total knee arthroplasty with patellar resurfacing.

DETAILED DESCRIPTION:
Anterior knee pain is an important cause of persistent pain after total knee arthroplasty. Lateral retinacular release has been proposed as a procedure to prevent anterior knee pain syndrome, based on the reduction of lateral tension and improving patellar tracking.

However, its effect on anterior knee pain after total knee arthroplasty is not clear when it is not strictly needed to correct maltracking.

The purpose of this trial is to evaluate the effect of systematic lateral retinaculare release on anterior knee pain, peformed during a total knee arthroplasty with patellar resurfacing.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of knee osteoarthritis

Exclusion Criteria:

* prior major surgery on the same knee (high tibial or distal femoral osteotomy, patellar realignment)
* important preoperative malalignment (varus or valgus >15º or flexion deformity >15º)
* inability to sign informed consent

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Anterior Knee Pain at one year after surgery | At the preoperative visit and at the 1-year follow up
  Pressure pain threshold determined using pressure algometry
Change from baseline in Knee Pain measured by Visual Analogue Scale at one year after surgery | At the preoperative visit and at the 1-year follow up
  The Visual Analogue Scale referred by the patients at rest, when walking and when going up and downstairs. Scored between 0 (no pain at all) and 10 (maximum pain the patient could imagine).

SECONDARY OUTCOMES:
Change from baseline in patellar pain and function at one year after surgery | At the preoperative visit and at the 1-year follow up
  Patellofemoral score designed by Feller, distributed with a maximum of 15 points for the intensity of anterior knee pain, 5 points for quadriceps strength, 5 points for the ability to rise from a chair and 5 points for stair climbing ability
Change from baseline in knee fuction, measured by the Knee Society Score, at one year after surgery | At the preoperative visit and at the 1-year follow up
  The Knee Society Score, being 0 the worst and 100 the best possible result

OTHER OUTCOMES:
Change from baseline in Patelar Height at one year after surgery | At the preoperative visit and at the 1-year follow up
  Measured in the lateral radiographic view using the Caton-Deschamps index
Change from baseline in Patellar Tilt at one year after surgery | At the preoperative visit and at the 1-year follow up
  Measured in the axial radiographic view, as the angle subtended by the anterior intercondylar line and the equatorial line of the patella preoperatively or a line drawn through the prosthesis-bone interface postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Parc de Salut Mar, Barcelona, Spain

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05778539/Prot_SAP_000.pdf